CLINICAL TRIAL: NCT00005241
Title: Myocardial Infarction and Current Oral Contraceptive Use
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1122; R01HL042483 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2001-06

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Myocardial Infarction; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Myocardial Infarction; Heart Diseases

SUMMARY:
To assess whether current oral contraceptive (OC) use (within the previous month) increased the risk of myocardial infarction. Also, to assess the combined effects of cigarette smoking and oral contraceptive use.

DETAILED DESCRIPTION:
BACKGROUND:

It has been established that oral contraceptive formulations used in the 1960s and 1970s increased the risks of myocardial infarction, venous thromboembolism, and stroke. Oral contraceptive formulations have changed, as have prescribing practices, and there was a need for information on the effects of the newer formulations in use. Myocardial infarction is the most important cardiovascular disease in terms of the incidence and mortality attributed to use of oral contraceptives; although the overall incidence of myocardial infarction is relatively low in women of childbearing ages, the incidence is not low in smokers.

DESIGN NARRATIVE:

A case-control design was used. The case series consisted of women 18 to 44 years of age admitted for a documented first myocardial infarction to any of 100 collaborating hospitals in Massachusetts, Rhode Island, and Pennsylvania. Nurse interviewers administered standard structured questionnaires to cases and controls on drug use, race, religion, medical history and myocardial infarction risk factors. Information was collected on: cigarette smoking; histories of hypertension, diabetes mellitus, angina, abnormal plasma lipids; reproductive and menstrual histories; alcohol and coffee consumption; personality type using the Framingham Type A scale; family history of myocardial infarction; exercise; education and occupation of the patient and her spouse. Information was also obtained on the timing and duration of oral contraceptive use. The effect of oral contraceptive use was considered among nonsmokers, light smokers, and heavy smokers. Individual oral contraceptive formulations were classified according to dosage and type of estrogen, formulation type, and other groupings. Multiple logistic regression analysis with fitting of the regression equations by the method of maximum likelihood was used for simultaneous control of all potential confounding factors.

The study was renewed in 1995 to continue data collection to establish the effect of triphasic OCs on MI risk, with particular attention to the joint effect with heavy smoking. The new data collection also permitted more definitive analysis of the effect of monophasic OCs. Triphasic formulations have become popular and in 1995 accounted for about half of OC use. There were not enough users of triphasic OCs in the present study for informative analysis, nor were there any data from other studies on this issue. The study ended in December, 1999.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-04; Study Completion 1999-12 (Actual)

REFERENCES:
- [Background] Rosenberg L, Palmer JR, Rao RS, Shapiro S. Low-dose oral contraceptive use and the risk of myocardial infarction. Arch Intern Med. 2001 Apr 23;161(8):1065-70. doi: 10.1001/archinte.161.8.1065. PMID 11322840